CLINICAL TRIAL: NCT03983057
Title: Study on Therapeutic Effect of Combination of Anti-PD-1 Antibody and Chemotherapy in Locally Advanced or Borderline Resectable Pancreatic Cancer Patients: A Randomized Clinical Trial
Brief Title: Combination of Anti-PD-1 Antibody and Chemotherapy in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISPD-4
Record Dates: First submitted 2019-06-05; First posted 2019-06-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; PD-1; FOLFIRINOX; combination therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy group (No Intervention): Treatment with modified-FOLFIRINOX Folic acid 400mg/m^2, 5- fluorouracil 2400mg/m^2 for 46h, irinotecan 135mg/m^2 and oxaliplatin 68mg/m^2
- Combination group (Experimental): Treatment with modified-FOLFIRINOX and Anti-PD-1 antibody Folic acid 400mg/m^2, 5- fluorouracil 2400mg/m^2 for 46h, irinotecan 135mg/m^2 and oxaliplatin 68mg/m^2, Anti-PD-1 antibody 3mg/kg
  Interventions: Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — Accompanying with modified-FOLFIRINOX, Anti-PD-1 antibody was applied biweekly.
  Arms: Combination group

SUMMARY:
The prognosis of pancreatic cancer is extremely poor. Current guidelines recommend FOLFIRINOX or modified-FOLFIRINOX as the first-line chemotherapeutic regimen. Studies have shown that immunotherapy with Anti-PD-1 antibody can effectively increase the response rate and prolong patient survival in a number of cancer diseases. Here investigators intend to compare the therapeutic effects of modified-FOLFIRINOX alone and the combination of modified-FOLFIRINOX and Anti-PD-1 antibody in patients with borderline resectable and locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Investigators chose borderline resectable and locally advanced pancreatic cancer patients. The planned treatment was given to the participants after randomization. Response rate, event-free survival, overall survival, drugs related side effects and other endpoints events were recorded and analyzed, to assess the combination treatment with modified-FOLFIRINOX and Anti-PD-1 antibody could or couldn't benefit the patients with borderline resectable and locally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed pancreatic ductal adenocarcinoma (PDAC).
* No evidence of distant metastasis (such as liver, peritoneum, lung) evaluated by abdominal contrast-enhanced CT, MRI, and chest CT. PET/CT or other imaging examinations would be used if necessary.
* Initial assessment for definitive borderline resectable or locally advanced tumors (resectability judgment is based on CT enhanced scan or magnetic resonance imaging, NCCN2019 first edition standard).
* ECOG score 0 or 1.
* Serum creatinine level is normal, and serum total bilirubin level is less than 1.5 x ULN.
* ALT and AST are less than 2 x ULN.
* If biliary obstruction is observed, biliary decompression should be performed when the patient is randomly assigned to receive neoadjuvant chemotherapy.
* Leukocyte count (> 3.5 x 10^6 /mL), neutrophil count (> 1.5 x 10^6 /mL), platelet count (> 80 x 10^6 /mL), hemoglobin (> 9 g/dL).
* Signed informed consent.

Exclusion Criteria:

* History of malignance treatment in the past, excluding basal and cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma
* History of participation of other clinical trails within 4 weeks
* History of immunotherapy within 4 weeks
* History of receiving chemotherapy, radiotherapy and molecular target therapy within 2 weeks
* Tumor is a local recurrent lesion.
* Imaging confirmed severe portal hypertension / cavernous transformation.
* Ascites
* Gastric outlet obstruction
* Respiratory failure requires supplementation of oxygen.
* Immune deficiency syndrome, such as active tuberculosis and HIV infection.
* Hematological precancerous diseases, such as myelodysplastic syndromes.
* Major cardiovascular diseases (including myocardial infarction, unstable angina, congestive heart failure, severe uncontrolled arrhythmia) during the past six months of enrollment.
* Evidence of clinical-related or previous interstitial lung disease, such as noninfectious pneumonia or pulmonary fibrosis, or baseline chest CT scan or chest X-ray findings
* Previous or physical findings of central nervous system disease, except for adequately treated (e.g. primary brain tumors, uncontrolled seizures or strokes with standard medications)
* Preexisting neuropathy > 1 (NCI CTCAE).
* Allograft requires immunosuppressive therapy or other major immunosuppressive therapies.
* Severe serious wounds, ulcers or fractures.
* Confirmed coagulant disease.
* Clinical evaluation is unacceptable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Event-free survival | From randomization to any of the following events: disease progression, local or distant recurrence, or death from any cause, whichever occurs first. Up to approximately 60 months.
  Event-Free Survival assessed by the investigator according to RECIST 1.1 by investigator, defined as the interval from randomization to the first occurrence of disease progression, local or distant recurrence, or death from any cause.

SECONDARY OUTCOMES:
Overall survival | From randomization to death due to any cause. Up to approximately 60 months.
  From randomization to death due to any cause.
Objective response rate | Up to approximately 60 months.
  The proportion of patients with tumor size reduction of a predefined amount and for a minimum time period
Disease control rate | Up to approximately 60 months.
  The proportion of patients with tumor size reduction or stable
Resection rate | Up to approximately 60 months.
  The proportion of patients with surgical treatment after treatment
R0 rate | Up to approximately 60 months.
  The proportion of patients with completely tumor resection after treatment
Adverse effects | Up to approximately 60 months.
  The most common hematologic and non-hemotologic adverse events
Carbohydrate antigen 19-9 | Up to approximately 60 months.
  Carbohydrate antigen 19-9 level

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No